CLINICAL TRIAL: NCT05896202
Title: Addressing Disparities in Neuromodulation for Rehabilitation: A Mixed Methods Approach to Optimize Access for Underrepresented Racial Minorities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Center of Neuromodulation for Rehabilitation (Other)
Responsible Party: Principal Investigator, Marlon Wong, Associate Professor of Clinical Physical Therapy, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20230154
Record Dates: First submitted 2023-05-31; First posted 2023-06-09 (Actual); Results first posted 2025-10-27 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Neuropathic Pain
Keywords: neurostimulation; video enhanced consent; neuromodulation; transcutaneous auricular vagus nerve stimulation; transcranial direct current stimulation; transcranial magnetic stimulation
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcutaneous Auricular Vagus Nerve stimulation (taVNS) group (Experimental): This group will receive supplemental videos on taVNS and TMS. Participants will be in this group for approximately 7 hours.
  Interventions: Other: taVNS Video; Other: Educational materials
- Transcranial Magnetic Stimulation (TMS) group (Active Comparator): This group will receive a supplemental video on TMS only. Participants will be in this group for approximately 7 hours.
  Interventions: Other: Educational materials; Other: TMS Video

INTERVENTIONS:
Other: taVNS Video — One third of the participants will see the taVNS video once in person. The video will be 2-3 minutes in length and contain information on the procedures of the technique and what participants should expect to feel/experience.
  Arms: Transcutaneous Auricular Vagus Nerve stimulation (taVNS) group
Other: Educational materials — Participants will receive sample consent forms and brochures for taVNS and TMS. These materials will be reviewed with each participant once on site, and they will have the opportunity to ask questions. participants will take these materials home and have the opportunity to review further at their leisure.
Other: TMS Video — One third of the participants will see the TMS video once in person. The video will be 2-3 minutes in length and contain information on the procedures of the technique and what participants should expect to feel/experience.
  Arms: Transcranial Magnetic Stimulation (TMS) group

SUMMARY:
The purpose of this study is to:

1. Development of culturally sensitive videos for enhance informed consent with neurostimulation and determination of factors that influence minority interest in participating in neurostimulation research.
2. Examination of the influence that video enhanced informed consent has on expectations with transcutaneous auricular vagus nerve stimulation (taVNS) and on treatment intended effects.

ELIGIBILITY:
Inclusion Criteria:

1. between the ages of 18-80 years
2. neuropathic pain lasting longer than 3 months (i.e., complaint of sensation of burning, stabbing or pressing pain, shooting or shock like pain, or paresthesias)
3. Neuropathic Pain Symptom Inventory score ≥10.
4. self identifies as Black or Hispanic

Exclusion Criteria:

1. any unstable medical condition or medical contraindication to moderate physical exertion (e.g., unstable angina or cardiac arrythmia)
2. pregnancy
3. currently taking Buprenorphine or recently stopped taking (within 1 month)
4. presence of cognitive impairment or language barrier that impairs full autonomy in the consent process or in the ability to participate in detailed interviews
5. implants in the head or neck, cochlear implants, or pacemaker
6. head or neck metastasis or recent ear trauma
7. history of seizures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-07-19 (Actual); Study Completion 2024-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marlon Wong, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wong ML, Widerstrom-Noga E, Bolanos JL, Gonzalez G, Penedo FJ, Hosein PJ, Tovin MM, Gonzalez JP, McTeague LM. Feasibility of trancutaneous auricular vagus nerve stimulation in Black and Hispanic/Latino people with peripheral neuropathy. Front Pain Res (Lausanne). 2025 Jan 17;5:1516196. doi: 10.3389/fpain.2024.1516196. eCollection 2024. PMID 39896735

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) Group | Transcranial Magnetic Stimulation (TMS) Group
Started | 14 | 14
Completed | 12 | 12
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) Group | Transcranial Magnetic Stimulation (TMS) Group | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (11.3) | 59.0 (7.5) | 58.6 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 5 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 8 | 18
  Not Hispanic or Latino | 4 | 6 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 9 | 16
  White | 6 | 5 | 11
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change Expectation for Pain Relief as Measured by EXPECT Scores
Description: The Expectations for Complementary and Alternative Medicine Treatments (EXPECT) is a 4-item questionnaire that assesses expectations for pain improvement. Each of the 4 items is scored on an 11-point scale, with 0 being no change and 10 representing complete relief (scores ranging from 0-10). Higher scores represent greater expectations for pain relief. Scores from all 4 items are summed to produce a total score ranging from 0 to 40, with higher scores indicating greater expectations for pain relief.
Time Frame: Baseline, and up to 90 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) Group | Transcranial Magnetic Stimulation (TMS) Group
Number analyzed (Participants) | 12 | 12
score on a scale | 0.19 (1.16) | 0.28 (1.08)

2. Secondary Outcome: Change in Heart Rate Variability (HRV)
Description: HRV will be measured with an H10 chest strap device measured in milliseconds (SDRR).
Time Frame: Baseline, up to 90 minutes
Measure: Mean (Standard Deviation); unit: Milliseconds
Groups:
- Active taVNS: Active stimulation applied to the cymba concha for 60 minutes
- Sham Stimulation: Active stimulation applied to the ear lobe for 60 minutes
Arm/Group | Active taVNS | Sham Stimulation
Number analyzed (Participants) | 11 | 11
Milliseconds | 0.42 (9.73) | -0.37 (12.89)

ADVERSE EVENTS:
Time Frame: 3 weeks
Arm/Group | Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) Group | Transcranial Magnetic Stimulation (TMS) Group
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-16): https://cdn.clinicaltrials.gov/large-docs/02/NCT05896202/Prot_SAP_000.pdf